CLINICAL TRIAL: NCT01074164
Title: Evaluating the Effectiveness of Acupressure in Relieving Pruritus Related to Atopic Dermatitis
Brief Title: Acupressure in Pruritus for Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Dennis West, Professor of Dermatology and Pediatrics, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 20535
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2013-01-16 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Atopic Dermatitis
Keywords: eczema; atopic dermatitis; itch; pruritus; acupressure; acupuncture
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): This group of subjects will serve as the control group and will follow a standard-of-care treatment regimen for AD, including the use of moisturizers and topical corticosteroids.
  Interventions: Other: Standard-of-care treatment for AD
- Accu-patch pellet (Experimental): This group of subjects will follow a standard-of-care treatment regimen for AD, including the use of moisturizers and topical corticosteroids. Additionally, they will use a titanium pellet (accu-patch pellet) to self-apply pressure at the LI11 acupuncture pressure point, located on the left arm lateral to the antecubital fossae, for 10 minutes, 3 times weekly for 1 month.
  Interventions: Device: Accu-patch pellet

INTERVENTIONS:
Other: Standard-of-care treatment for AD — Subjects will receive standard of care treatment for atopic dermatitis, including moisturizers and topical corticosteroids, per their dermatologist.
  Arms: Control group
Device: Accu-patch pellet — The accu-patch pellets will be applied to the LI11 pressure point, located on the left arm lateral to the antecubital fossae, for 10 minutes, 3 times a week for 1 month.
  Arms: Accu-patch pellet

SUMMARY:
The purpose of this study is to see if acupressure will be effective at reducing itch in people with atopic dermatitis (AD).

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is recognized as a major and common problem worldwide. In the United States, AD and related eczematous symptoms affect 17% of the population; 1 in 10 individuals report having experienced symptoms causing quality of life (QOL) distress, including itching/scratching, red/inflamed rash, excessive dryness/scaling, and/or symptoms lasting ≥ 14 days. Two-thirds of these subjects noted at least moderate to severe symptoms, with itch being the most disturbing. Effective treatment of AD and of pruritus (itching) are interconnected. Treating AD will decrease the stimulus for the itch, whereas treating pruritus will decrease the feedback cycle brought on when a patient scratches the skin continually. Effective medications for AD and related symptoms include topical corticosteroids and calcineurin inhibitors. Oftentimes, these remedies are insufficient at treating the itch component of the disease. There is demand for alternative, complementary treatments for AD-related pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD by dermatologist
* Not currently using acupressure or acupuncture for treatment of AD
* Able to read, write, and understand study materials
* Age 18 or older

Exclusion Criteria:

* Unable to physically perform acupressure technique
* Significant comorbidities causing itch such as chronic urticaria, renal failure, notalgia paresthetica, and tinea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis West, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: This group of subjects served as the control group and followed a standard-of-care treatment regimen for AD, including the use of moisturizers and topical corticosteroids.
- Accu-patch Pellet: This group of subjects followed a standard-of-care treatment regimen for AD, including the use of moisturizers and topical corticosteroids. Additionally, they used a titanium pellet (accu-patch pellet) to self-apply pressure at the LI11 acupuncture pressure point, located on the left arm lateral to the antecubital fossae, for 10 minutes, 3 times weekly for 1 month.
Period: Overall Study
Arm/Group | Control Group | Accu-patch Pellet
Started | 7 | 8
Completed | 4 | 7
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Accu-patch Pellet | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (18.3) | 35.1 (11.3) | 37.3 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Itch Intensity as Measured by a Change in Visual Analog Scale (VAS) Score
Description: The VAS score assesses itch intensity in subject's with AD. The VAS consists of a 21.5 cm horizontal line with its left and right boundaries marked by vertical lines. The left boundary vertical line is labeled "Least Itch," and the right boundary vertical line is labeled "Worst Itch." Subjects are instructed to draw a vertical line across this scale that represents the intensity of itch that they are currently experiencing. Vertical lines drawn by subjects towards the left boundary of the horizontal line are associated with less itch intensity, and vertical lines drawn by subjects towards the right boundary of the horizontal line are associated with worse itch intensity. A ruler is then used to measure distance from the left boundary vertical line to the vertical line drawn by the subject to the nearest millimeter. Possible values range from 0 to 21.5 centimeters, with 0 centimeters associated with less itch intensity and 21.5 cm associated with worse itch intensity.
Time Frame: Baseline and 4 weeks
Measure: Mean (Full Range); unit: centimeters
Arm/Group | Control Group | Accu-patch Pellet
Number analyzed (Participants) | 4 | 7
centimeters | 0.8 [-3.2 to 1.8] | -5.0 [-11.0 to 0.5]

2. Secondary Outcome: Change in Severity of Atopic Dermatitis (AD) as Measured by a Change in Investigator Global Assessment (IGA) Score
Description: The IGA score is an assessment of AD severity. It is an assessment of the patient's disease state at the time of examination and does not attempt a comparison with any of the patient's previous disease states. Possible scores range from 0 to 5. A score of 0 is associated with no evidence of AD and a score of 5 is associated with severe AD.
Time Frame: Baseline and 4 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control Group | Accu-patch Pellet
Number analyzed (Participants) | 4 | 7
units on a scale | 0.5 [0 to 3] | -1 [-3 to 0]

3. Secondary Outcome: Change in Severity of Atopic Dermatitis (AD) as Measured by a Change in Eczema Area and Severity Index (EASI): Area Subscale Score
Description: The EASI is a composite score assessing four key clinical signs of AD and the area of skin involvement in four main body regions (head, trunk, upper limbs, and lower limbs). The 5 EASI subscales are: erythema, infiltration/papulation, excoriation, lichenification, and percent area of skin involvement. For determining area subscale score, the percent area of skin involvement is determined and assigned a score of 0 to 6, where 0 correlates with no skin involvement, 1 represents < 10% skin involvement, 2 represents 10-29% skin involvement, 3 represents 30-49% skin involvement, 4 represents 50-69% skin involvement, 5 represents 70-89% skin involvement, and 6 represents 90-100% skin involvement. Possible scores range from 0 to 6, where 0 correlates with better disease severity and 6 correlates with worse disease severity.
  Hanifin JM, Thurston M, Omoto M, et al (2001) The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. Exp Dermatol; 10: 11-18.
Time Frame: Baseline and 4 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Control Group | Accu-patch Pellet
Number analyzed (Participants) | 4 | 7
units on a scale | 0 [0 to 1] | -1 [-3 to 1]

4. Secondary Outcome: Change in Severity of Atopic Dermatitis (AD) as Measured by a Change in Eczema Area and Severity Index (EASI): Erythema Subscale Score
Description: The EASI is a composite score assessing four key clinical signs of AD and the area of skin involvement in four main body regions (head, trunk, upper limbs, and lower limbs). The 5 EASI subscales are: erythema, infiltration/papulation, excoriation, lichenification, and percent area of skin involvement. For determining the erythema subscale score, erythema is assessed in each main body region and assigned a score of 0 to 3, where a score of 0 is associated with no expression of the clinical sign and a score of 3 is associated with severe expression of the clinical sign. Possible scores range from 0 to 3, where 0 correlates with better disease severity and 3 correlates with worse disease severity.
  Hanifin JM, Thurston M, Omoto M, et al (2001) The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. Exp Dermatol; 10: 11-18.
Time Frame: Baseline and 4 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Control Group | Accu-patch Pellet
Number analyzed (Participants) | 4 | 7
units on a scale | 0 [-1 to 1] | -1 [-3 to 1]

5. Secondary Outcome: Change in Severity of Atopic Dermatitis (AD) as Measured by a Change in Eczema Area and Severity Index (EASI): Infiltration/Papulation Subscale Score
Description: The EASI is a composite score assessing four key clinical signs of AD and the area of skin involvement in four main body regions (head, trunk, upper limbs, and lower limbs). The 5 EASI subscales are: erythema, infiltration/papulation, excoriation, lichenification, and percent area of skin involvement. For determining the infiltration/papulation subscale score, infiltration/papulation is assessed in each main body region and assigned a score of 0 to 3, where a score of 0 is associated with no expression of the clinical sign and a score of 3 is associated with severe expression of the clinical sign. Possible scores range from 0 to 3, where 0 correlates with better disease severity and 3 correlates with worse disease severity.
  Hanifin JM, Thurston M, Omoto M, et al (2001) The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. Exp Dermatol; 10: 11-18.
Time Frame: Baseline and 4 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Control Group | Accu-patch Pellet
Number analyzed (Participants) | 4 | 7
units on a scale | 0 [-2 to 1] | -1 [-2 to 0]

6. Secondary Outcome: Change in Severity of Atopic Dermatitis (AD) as Measured by a Change in Eczema Area and Severity Index (EASI): Excoriation Subscale Score
Description: The EASI is a composite score assessing four key clinical signs of AD and the area of skin involvement in four main body regions (head, trunk, upper limbs, and lower limbs). The 5 EASI subscales are: erythema, infiltration/papulation, excoriation, lichenification, and percent area of skin involvement. For determining the excoriation subscale score, excoriation is assessed in each main body region and assigned a score of 0 to 3, where a score of 0 is associated with no expression of the clinical sign and a score of 3 is associated with severe expression of the clinical sign. Possible scores range from 0 to 3, where 0 correlates with better disease severity and 3 correlates with worse disease severity.
  Hanifin JM, Thurston M, Omoto M, et al (2001) The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. Exp Dermatol; 10: 11-18.
Time Frame: Baseline and 4 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Control Group | Accu-patch Pellet
Number analyzed (Participants) | 4 | 7
units on a scale | 0 [-2 to 2] | -1 [-2 to 0]

7. Secondary Outcome: Change in Severity of Atopic Dermatitis (AD) as Measured by a Change in Eczema Area and Severity Index (EASI): Lichenification Subscale Score
Description: The EASI is a composite score assessing four key clinical signs of AD and the area of skin involvement in four main body regions (head, trunk, upper limbs, and lower limbs). The 5 EASI subscales are: erythema, infiltration/papulation, excoriation, lichenification, and percent area of skin involvement. For determining the lichenification subscale score, lichenification is assessed in each main body region and assigned a score of 0 to 3, where a score of 0 is associated with no expression of the clinical sign and a score of 3 is associated with severe expression of the clinical sign. Possible scores range from 0 to 3, where 0 correlates with better disease severity and 3 correlates with worse disease severity.
  Hanifin JM, Thurston M, Omoto M, et al (2001) The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. Exp Dermatol; 10: 11-18.
Time Frame: Baseline and 4 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Control Group | Accu-patch Pellet
Number analyzed (Participants) | 4 | 7
units on a scale | 0 [-1 to 1] | -1 [-2 to 0]

ADVERSE EVENTS:
Arm/Group | Control Group | Accu-patch Pellet
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes